CLINICAL TRIAL: NCT03560388
Title: Assessing Effectiveness of Acupuncture and Integrative Care in Reducing Peri- and Intra-operative Pain and Anxiety in Patients With Gynecological Cancer: A Randomized Controlled Study
Brief Title: Acupuncture and Integrative Care in Gynecological Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Eran Ben-Arye, Clinical Associate Professor, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CMC-18-0037-CTIL
Record Dates: First submitted 2018-05-02; First posted 2018-06-18 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Quality of Life
Keywords: Integrative medicine; Acupuncture; Gynecological oncology; Surgery; Analgesia; Pain; Anxiety
MeSH Terms: conditions — Agnosia; Pain; Anxiety Disorders | interventions — Acupuncture Therapy; Touch

STUDY DESIGN:
Intervention Model Description: Two main arms of control and intervention. Intervention arm include two sub-arms of integrative treatment plus acupuncture vs. integrative treatment with no acupuncture
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participant, care provider, and investigator are blind to allocation to control vs. intervention groups. Participant is also blind to the 2nd allocation to the two intervention group sub-arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Control group include participants randomly allocated to supportive care (with no added integrative care or acupuncture)
- Touch/relaxation (Experimental): Touch/relaxation treatment (pre-operative)
  Interventions: Other: Acupuncture and touch/relaxation
- Acupuncture and touch/relaxation (Experimental): Acupuncture (intra operative) and touch-relaxation treatment (pre-operative)
  Interventions: Other: Acupuncture and touch/relaxation

INTERVENTIONS:
Other: Acupuncture and touch/relaxation — Pre-operative integrative care (touch-relaxation) that follows with intra-operative acupuncture
  Arms: Acupuncture and touch/relaxation; Touch/relaxation

SUMMARY:
Patients undergoing surgical procedures for gynecological cancer are frequently challenged by intense anxiety prior to surgery, reflecting the accompanying uncertainty regarding the diagnosis, treatment and prognosis of their illness.The purpose of the proposed study is to explore the impact of complementary and integrative medicine (CIM) treatments (including acupuncture) on anxiety, pain, and general QOL of patients referred to gynecological oncology surgery. The investigators working hypothesis is that an intensive CIM treatment program, provided to patients within 24 hours prior to and during surgery will reduce perioperative anxiety and pain, and will reduce the need for intra-operative and post-operative analgesia.

DETAILED DESCRIPTION:
Patients undergoing surgical procedures for gynecological cancer are frequently challenged by intense anxiety prior to surgery, reflecting the accompanying uncertainty regarding the diagnosis, treatment and prognosis of their illness. Following operation, pain and other quality of life-related concerns further exacerbate the emotional distress, which may itself aggravate pain and other symptoms. Clinical, controlled studied among patients with gynecological cancer undergoing chemotherapy had demonstrated effectiveness of complementary and integrative medicine (CIM) treatments for improving quality of life (QOL) and related symptoms, such as pain, gastro-intestinal concerns, fatigue, and anxiety.

The purpose of the proposed study is to explore the impact of CIM treatments (including acupuncture) on anxiety, pain, and general QOL of patients referred to gynecological oncology surgery. The investigators' working hypothesis is that an intensive CIM treatment program, provided to patients within 24 hours prior to and during surgery will reduce perioperative anxiety and pain, and will reduce the need for intra-operative and post-operative analgesia.

ELIGIBILITY:
Inclusion Criteria: Female patients age ≥ 18 years, who were referred to surgery for suspected/established gynecological-oncology cancer at the Carmel Medical Center; Patients diagnosed with class1-3 peri-operative risk according to American Society of Anesthesia.

Exclusion Criteria:Unwillingness to sign the research participation form and/or limitations in comprehending the informed consent; during pregnancy; patients with chronic pain treated with opiates within one month preceding surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients undergoing gynecologic-oncology surgery
Enrollment: 135 (Estimated)
Dates: Start 2018-06-24 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain assessment change | Change from pre- (1 hour before) to post-operative (24 hours following surgery)
  Pain assessment on a visual analogue scale

SECONDARY OUTCOMES:
Anxiety assessment change | Change from pre- (1 hour before) to post-operative (24 hours following surgery)
  Anxiety assessment on a visual analogue scale
Reduced analgesics use | During surgery (4-6 hours) and 24-hour post-surgery
  Monitoring intra- and post-operative analgesia use

CONTACTS AND LOCATIONS:
Overall Officials: Eran Ben-Arye, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Carmel Medical center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Segev Y, Abofol S, Samuels N, Schmidt M, Assaf W, Ben-Arye E. Postoperative pain following intraoperative acupuncture: a randomized-controlled study. BMJ Support Palliat Care. 2025 Aug 26;15(5):642-647. doi: 10.1136/spcare-2025-005485. PMID 40537176